CLINICAL TRIAL: NCT06863857
Title: Dual-energy SPEctral CT to Evaluate Response to New First-line Therapies in Patients With Metastatic Clear Cell REnal Cancer and the Association of Its Parameters With Molecular Alterations
Brief Title: Dual-energy SPEctral CT to Evaluate Response to First-line Therapies in Patients With Metastatic Clear Cell REnal Cancer
Acronym: SPECTRE
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: SPECTRE
Record Dates: First submitted 2025-01-10; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2024-11

CONDITIONS: Renal Cancer
Keywords: Dual energy spectral CT
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Tissue sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the utility of dual-energy spectral computed tomography (CT) scan in monitoring treatment in patients with metastatic clear cell carcinoma of the kidney. In particular, to analyze the use of spectral CT in patients who are candidates to receive first-line treatment based on combinations of immunotherapy and molecularly targeted drugs. In particular, the parameters derived from the use of this technology and their variation during therapy will be analyzed together with some possible molecular alterations highlighted by the analysis of the tumor tissue previously taken from the patient, relating them to the response to first-line therapy with immuno-combinations.

DETAILED DESCRIPTION:
In the field of kidney cancer, where PET with FDG or other tracers is not valid due to the high number of false negatives, new techniques for radiological evaluation of the disease are a clinical necessity. The evaluation of parameters derived from the use of dual-energy spectral computed tomography (CT), such as IC and Zeffective, at baseline and after 3 and 6 months of systemic treatment, could provide useful information on how tumor structure (in particular vascularization) evolves during therapy with IO+IO or IO+TKI. In addition, the variation of these parameters could be associated with different outcomes in terms of ORR, PFS and OS. One aspect evaluated is the existence of a correlation between the presence of abundant tumor vascularization (or on the contrary poor vascularization), determined by dual-energy spectral CT, and the response in terms of ORR and PFS at 3 and 6 months to combinations containing IO+TKI or immunotherapy alone. For prognostic and predictive purposes, the study also intends to verify whether there is a correlation between the presence of gene alterations, CT-derived parameters and response to therapies. The prognostic role of some molecular alterations (ATM, BAP1, KDM5C, MET, MTOR, NF2, PBRM1, PIK3CA, PTEN, SETD2, SMARCB1, TP53, TSC1, TSC2, VHL) will be evaluated and their potential predictive value will be analyzed to understand whether a given mutational structure may be more or less responsive to specific types of treatment.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years
* Patients with histological or cytological diagnosis of clear cell RCC
* Patients with metastatic disease documented by imaging or biopsy of the secondary site
* Patients who have not had previous treatment for RCC
* Patients with an indication for first-line medical treatment based on IO+TKI, IO+IO as per clinical practice at the Medical Oncology Unit of the IRCCS University Hospital of Bologna
* Patients who have already had a dual-energy spectral total-body CT with MDC within 4 weeks of treatment initiation
* Availability of a formalin-fixed, paraffin-embedded histological block (FFPE) stored for a period <15 years, for the execution of molecular analysis for the search for alterations of the genes ATM, BAP1, KDM5C, MET, MTOR, NF2, PBRM1, PIK3CA, PTEN, SETD2, SMARCB1, TP53, TSC1, TSC2, VHL
* Patients who knowingly express consent to participate in the study after signing the consent

Exclusion Criteria

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients diagnosed with metastatic ccRCC and who comply with study inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2027-06-18 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Response to first-line drug therapy (with immuno-combinations) in patients with metastatic renal cell carcinoma | From enrollment to 6 months of systemic therapy
  IC and Zeffective parameters will be compared between responders and non-responders. the outcome studied will be the Overall Response Rate (ORR) assessed radiologically according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Overall Survival (OS) | From enrollment to 12 months of sistemic therapy
  for prognostic value of dual-energy spectral CT-derived parameters: Overall Survival (OS) at 12 months For prognostic impact of molecular alterations: OS at 12 months after initiation of therapy.
Progression-free survival (PFS) | From enrollment to 6 months of sistemic therapy
  for prognostic value of dual-energy spectral CT-derived parameters: Overall Survival (OS) at 12 months and Progression-Free Survival (PFS) at 6 months after initiation of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Massari, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- Italy (2):
  - Irccs Azienda Ospedaliero Universitario Di Bologna, Bologna, BO
  - Oncology Unit, IRCCS Azienda Ospedaliero Universitaria Bologna, Bologna

IPD SHARING:
Plan to Share IPD: No